CLINICAL TRIAL: NCT05271968
Title: Place of Hygiene in Scabies's Treatment in Populations in Precarious Situations
Acronym: GALEHYGIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP210864
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Scabies
Keywords: Contagious disease; Scabies infection; Poor condition; Hygiene
MeSH Terms: conditions — Scabies; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard Care : The classic treatment recommended is the prescription of an oral drug, Ivermectin to be taken two times at one or 2 weeks interval. And recommendations on the need to change the clothes and the linen of the bedding the following day after taking the drug, washing them at more than 50° as well as all the clothes three days before are explained. The first course of oral treatment is swallowed at the BOPC, while the second course is given to be swallowed one week later.
- Intervention (Experimental): Patients in this interventional arm will come back to BOPC the following day after intake the treatment (D1 and D8) to take a shower and to receive again new clothes
  Interventions: Procedure: Global management of scabies

INTERVENTIONS:
Procedure: Global management of scabies — For the interventional arm, the first course of the oral treatment has also to be swallowed at the BOPC service, but the patient will have to come back the following day to take a shower at the BOPC service and will receive new clothes.
  The second course will be given, but the patient will have to come back the following day of the second course to take a shower at the BOPC service and to receive again new clothes
  Arms: Intervention

SUMMARY:
Scabies is a parasitic pathology contracted mainly through human contamination. It is caused by a parasite (Sarcoptes Scabiei var. hominis) which lodges into the top layer of the epidermis creating a burrow, which can measure 5 mm to 15 mm, where the female lays her eggs.

After 4-6 weeks the patient develops an allergic reaction to the presence of mite proteins and feces in the scabies burrow, causing intense itch and rash. The usual adult form, called common scabies, is characterized by this nocturnal pruritus, and typical and/or atypical lesions. The typical lesions are the vesicle (translucent vesicle on an erythematous base), the scabious burrow (due to the tunnel dug by the female in the stratum), and the papulo- nodule -nodular scabious (red/brown infiltrated on palpation, predominantly on the male genital areas). They predominate in certain regions: the interdigital region of the hands, the anterior face of the wrists, the external face of the elbows, the axillary region, the areolas, the nipples, the umbilical region, the male external genitalia, the buttock region, the face inner thighs.

Scabies occurs worldwide. However, studies have shown a greater prevalence among populations that do not have access to common hygiene measures: poor, young children and elderly in resource -poor communities, migrant, homeless populations, etc. The "Baudelaire outpatient clinic" (BOPC) at St Antoine hospital in Paris offers general medicine consultations. It has the particularity of offering a so called "Permanent d'Accès Aux Soins" service that allowed any person without health assurance to have access to a general practitioner and treatment, free of charge and help to recover its social rights. Consequently, more than 60% of the patients encountered at the consultation of the BOPC are in a precarious situation.

Usually, poor patients with scabies may be offered a shower and clean clothes at the BOPC Therefore it seemed to us the ideal place to evaluate a treatment's scabies in this population including the hygiene treatment.

DETAILED DESCRIPTION:
The objective of our study is to evaluate the superiority of a global management of scabies compared to a conventional treatment.

The classic treatment recommended is the prescription of an oral drug, Ivermectin to be taken two times at one or 2 weeks interval. And recommendations on the need to change the clothes and the linen of the bedding the following day after taking the drug, washing them at more than 50° as well as all the clothes three days before are explained. The first course of oral treatment is swallowed at the BOPC, while the second course is given to be swallowed one week later.

For the interventional arm, the first course of the oral treatment has also to be swallowed at the BOPC but the patient will have to come back the following day to take a shower at the BOPC and will receive new clothes. The second course will be given, but the patient will have to come back the following day of the second course to take a shower at the BOPC and to receive again new clothes.

We will compare the number of patients cured in the interventional arm versus the control arm at D28.

ELIGIBILITY:
Inclusion Criteria:

* Patient seen in consultation at the outpatient clinic, diagnosed with non-hyperkeratotic scabies.
* Living on the streets or without access to body care.
* Having received information on the protocol and having signed consent

Exclusion Criteria :

* Patient alcoholic on the day of the consultation
* Medical history fo psychiatric disease , severe somatic comorbidity, allergy to Ivermectin, pregnant woman
* Patient not understanding the on-site management (shower, change of clothes, taking the first dose of the drug on site)
* Non-communicating patient
* Hyperkeratotic or impetiginized scabies
* Patients not reachable by phone
* Patient having been treated for scabies less than 45 days before
* Patients under guardianship / curator ship or adults and subject to another protective measure.
* Pregnant and breastfeeding women
* Persons deprived of liberty by judicial and administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Healing | 28 days
  To assess the impact on the scabies healing rate by providing to patient in precarious situation a shower and clean clothes, twice at one-week intervals, versus the standard hygiene recommendations given to patients.
  Number of patients cured in the interventional arm (P=Policlinic) versus the control arm (D=home) at D28.

SECONDARY OUTCOMES:
Compliance | 28 days
  Compliance with treatment and effectiveness of the proposed device: determination of the number of patients seen again on D2 and D8 for the shower, and on D28 for the two groups.
Validity of the proposed clinical criteria | 28 days
  Validity of the proposed clinical criteria: the cure rate in each group will be analyzed according to the three clinical grades, confirmed, probable and possible

CONTACTS AND LOCATIONS:
Overall Officials: Bacha Kaoutar, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Saint Antoine - Polyclinique Beaudelaire, Paris, Ap-hp, France